CLINICAL TRIAL: NCT05408689
Title: A Randomized Controlled Clinical Trial of Transcutaneous Electrical Nerve Stimulation to Improve the Cognitive Functions in Older Adults
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) to Improve the Cognitive Functions in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022_TVNS
Record Dates: First submitted 2022-05-29; First posted 2022-06-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive function; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T1 TENS (Experimental): In this study, participants will be treated 30 min per day, 3 days per week, for 10 consecutive weeks
  Interventions: Device: T1 TENS
- Concha TENS (Experimental): In this study, participants will be treated 30 min per day, 3 days per week, for 10 consecutive weeks
  Interventions: Device: Concha TENS
- Control (Placebo Comparator): In this study, participants will be treated 30 min per day, 3 days per week, for 10 consecutive weeks
  Interventions: Device: Control

INTERVENTIONS:
Device: T1 TENS — The subjects in Group A will received TENS (Burst mode, 9 pulses per burst, pulse frequency =160Hz, burst frequency=2Hz, intensity was set to trigger visible muscular twitches). Two 2 x 3 cm electrodes was attached on T1 level with 2 cm from the spine. Previous study has shown that it was effective to improve the cognitive function in subjects with Alzheimer's disease.
  Arms: T1 TENS
Device: Concha TENS — The subjects in Group B will received TENS (25Hz, 0.5mA) on the concha of left outer ear. The electrical stimulation was generated by the portable neurostimulator (Nemos®, Cerbomed, Erlangen, Germany) and was delivered by a titanium electrodes positioning on top of a silicon earplug. Previous study has shown that it was effective to improve the Accelerate extinction memory formation and retention in healthy young adults.
  Arms: Concha TENS
Device: Control — The subjects in Group C will receive 30 min sham electrical stimulation on T1 by a placebo-TENS device. The Placebo-TENS was applied by an apparently identical TENS unit. The unit's power indicator light was illuminated, but the unit's electrical circuit had been manually disconnected inside. In order to shape the common mindset, all subjects (except those in the Control group) were informed that they might or might not feel an electrical current, as different stimulation parameters were being applied.
  Arms: Control

SUMMARY:
Recent evidence has shown that transcutaneous electrical nerve stimulation (TENS) was effective in improving the cognitive function in healthy adult and people with dementia. However, lacking of evidence investigated the effect of TENS in improving the cognitive function and reversing the occurrence of dementia during the period of mild cognitive impairment (MCI), which is the crucial period to prevent the significant loss of cognition function. Therefore, the main objective of this study is to investigate the optimal TENS treatment protocol in improving the cognitive function in older adults with MCI.

DETAILED DESCRIPTION:
This study aims to investigate the effectiveness of 3 intervention protocols (1) In the T1 TENS group, the subject will receive TENS on T1 spine. (2) In the vagus nerve TENS group, the subject will receive TENS on the concha of left outer ear. (3) In the sham stimulation group, the subject will receive sham stimulation on the T1 spine, in improving the cognitive function in older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

Should fulfil the diagnosis criteria of MCI (Albert et al., 2011):

1. Concern regarding a change in cognition
2. Impairment in one or more cognitive domains
3. Preservation of independence in functional abilities
4. no signs of dementia were to be present and confirmed by the medical staff and medical records.

Exclusion Criteria:

1. If their medical records reported a history of either psychiatric disorder, alcoholism, cerebral trauma, cerebrovascular disease, hydrocephalus, neoplasm, epilepsy, disturbances of consciousness, insulin-dependent diabetes mellitus or focal brain disorders;
2. Having active implants, such as cochlear implants, pacemaker;
3. Having wounds and diseased skin on the electrode position.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Montreal cognitive assessment (MoCA) | Baseline (0 week)
  The overall cognitive function is measured by the Cantonese version of MoCA. The MoCA is a widely used 10-minute cognitive screening test for detection of MCI. The MoCA test includes 8 parts with a maximum score of 30. A higher score indicated a better cognitive function. The Cantonese version of MoCA has shown good to excellent inter-rater (ICC=0.987, p<0.001) reliability in Chinese older adults.
Montreal cognitive assessment (MoCA) | Mid-intervention (5 week)
  The overall cognitive function is measured by the Cantonese version of MoCA. The MoCA is a widely used 10-minute cognitive screening test for detection of MCI. The MoCA test includes 8 parts with a maximum score of 30. A higher score indicated a better cognitive function. The Cantonese version of MoCA has shown good to excellent inter-rater (ICC=0.987, p<0.001) reliability in Chinese older adults.
Montreal cognitive assessment (MoCA) | Post-intervention (10 week)
  The overall cognitive function is measured by the Cantonese version of MoCA. The MoCA is a widely used 10-minute cognitive screening test for detection of MCI. The MoCA test includes 8 parts with a maximum score of 30. A higher score indicated a better cognitive function. The Cantonese version of MoCA has shown good to excellent inter-rater (ICC=0.987, p<0.001) reliability in Chinese older adults.
Montreal cognitive assessment (MoCA) | 1 month follow-up (14 week)
  The overall cognitive function is measured by the Cantonese version of MoCA. The MoCA is a widely used 10-minute cognitive screening test for detection of MCI. The MoCA test includes 8 parts with a maximum score of 30. A higher score indicated a better cognitive function. The Cantonese version of MoCA has shown good to excellent inter-rater (ICC=0.987, p<0.001) reliability in Chinese older adults.
Digit Span Test | Baseline (0 week)
  The verbal short-term memory and working memory is measured by the digit span test. The subject was required to listen to a series of random numbers carefully and then repeated them in forward (forward digit span test) and backward (backward digit span test) order. Continue in the same manner by increasing the series of numbers. The difficulty will be increased when the number in a sequence increased. The forward digit span task requires verbal working memory and attention, while the backwards digit span task additionally tests cognitive control and executive function. The more correct trials performed indicated better short-term memory and work memory.
Digit Span Test | Mid-intervention (5 week)
  The verbal short-term memory and working memory is measured by the digit span test . The subject was required to listen to a series of random numbers carefully and then repeated them in forward (forward digit span test) and backward (backward digit span test) order. Continue in the same manner by increasing the series of numbers. The difficulty will be increased when the number in a sequence increased. The forward digit span task requires verbal working memory and attention, while the backwards digit span task additionally tests cognitive control and executive function.The more correct trials performed indicated better short-term memory and work memory.
Digit Span Test | Post-intervention (10 week)
  The verbal short-term memory and working memory is measured by the digit span test. The subject was required to listen to a series of random numbers carefully and then repeated them in forward (forward digit span test) and backward (backward digit span test) order. Continue in the same manner by increasing the series of numbers. The difficulty will be increased when the number in a sequence increased. The forward digit span task requires verbal working memory and attention, while the backwards digit span task additionally tests cognitive control and executive function.The more correct trials performed indicated better short-term memory and work memory.
Digit Span Test | 1 month follow-up (14 week)
  The verbal short-term memory and working memory is measured by the digit span test . The subject was required to listen to a series of random numbers carefully and then repeated them in forward (forward digit span test) and backward (backward digit span test) order. Continue in the same manner by increasing the series of numbers. The difficulty will be increased when the number in a sequence increased. The forward digit span task requires verbal working memory and attention, while the backwards digit span task additionally tests cognitive control and executive function.The more correct trials performed indicated better short-term memory and work memory.
Visual Memory Span Test | Baseline (0 week)
  The visual memory is measured by the visual memory span test. The subject was required to observe a given order to tap a number of block as shown by the examiners and then repeat them in forward and backward order. The difficulty will be increased when the number of blocks in a sequence increased. The more correct trials performed indicated better visual memory.
Visual Memory Span Test | Mid-intervention (5 week)
  The visual memory is measured by the visual memory span test. The subject was required to observe a given order to tap a number of block as shown by the examiners and then repeat them in forward and backward order. The difficulty will be increased when the number of blocks in a sequence increased. The more correct trials performed indicated better visual memory.
Visual Memory Span Test | Post-intervention (10 week)
  The visual memory is measured by the visual memory span test. The subject was required to observe a given order to tap a number of block as shown by the examiners and then repeat them in forward and backward order. The difficulty will be increased when the number of blocks in a sequence increased. The more correct trials performed indicated better visual memory.
Visual Memory Span Test | 1 month follow-up (14 week)
  The visual memory is measured by the visual memory span test. The subject was required to observe a given order to tap a number of block as shown by the examiners and then repeat them in forward and backward order. The difficulty will be increased when the number of blocks in a sequence increased. The more correct trials performed indicated better visual memory.
Stroop Color and Word Test | Baseline (0 week)
  The ability to inhibit cognitive interference is measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Stroop Color and Word Test | Mid-intervention (5 week)
  The ability to inhibit cognitive interference is measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Stroop Color and Word Test | Post-intervention (10 week)
  The ability to inhibit cognitive interference is measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Stroop Color and Word Test | 1 month follow-up (14 week)
  The ability to inhibit cognitive interference is measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Face Recognition Test | Baseline (0 week)
  The visual, nonverbal long-term memory is measured by the face recognition test from the Rivermead Behavioral Memory Test (RMBT). Fifteen faces are shown successively to the subject. After an occupied interval of 5 minutes, the subjects are required to select the original 15 faces from a set of 30. The recognition score is the number of correct answers minus the number of incorrect answers. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, nonverbal long term memory.
Face Recognition Test | Mid-intervention (5 week)
  The visual, nonverbal long-term memory is measured by the face recognition test from the Rivermead Behavioral Memory Test (RMBT). Fifteen faces are shown successively to the subject. After an occupied interval of 5 minutes, the subjects are required to select the original 15 faces from a set of 30. The recognition score is the number of correct answers minus the number of incorrect answers. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, nonverbal long term memory.
Face Recognition Test | Post-intervention (10 week)
  The visual, nonverbal long-term memory is measured by the face recognition test from the Rivermead Behavioral Memory Test (RMBT). Fifteen faces are shown successively to the subject. After an occupied interval of 5 minutes, the subjects are required to select the original 15 faces from a set of 30. The recognition score is the number of correct answers minus the number of incorrect answers. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, nonverbal long term memory.
Face Recognition Test | 1 month follow-up (14 week)
  The visual, nonverbal long-term memory is measured by the face recognition test from the Rivermead Behavioral Memory Test (RMBT). Fifteen faces are shown successively to the subject. After an occupied interval of 5 minutes, the subjects are required to select the original 15 faces from a set of 30. The recognition score is the number of correct answers minus the number of incorrect answers. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, nonverbal long term memory.
Picture Recognition Test | Baseline (0 week)
  The visual, verbal long-term memory is measured by the picture recognition test from the RBMT. Line drawings of 15 common objects are presented one at a time. After an occupied interval of 5 minutes, the subjects are asked to select the original 15 pictures from a set of 30. The recognition score is calculated in the same way as in the Face Recognition test. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, verbal long term memory.
Picture Recognition Test | Mid-intervention (5 week)
  The visual, verbal long-term memory is measured by the picture recognition test from the RBMT. Line drawings of 15 common objects are presented one at a time. After an occupied interval of 5 minutes, the subjects are asked to select the original 15 pictures from a set of 30. The recognition score is calculated in the same way as in the Face Recognition test. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, verbal long term memory.
Picture Recognition Test | Post-intervention (10 week)
  The visual, verbal long-term memory is measured by the picture recognition test from the RBMT. Line drawings of 15 common objects are presented one at a time. After an occupied interval of 5 minutes, the subjects are asked to select the original 15 pictures from a set of 30. The recognition score is calculated in the same way as in the Face Recognition test. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, verbal long term memory.
Picture Recognition Test | 1 month follow-up (14 week)
  The visual, verbal long-term memory is measured by the picture recognition test from the RBMT. Line drawings of 15 common objects are presented one at a time. After an occupied interval of 5 minutes, the subjects are asked to select the original 15 pictures from a set of 30. The recognition score is calculated in the same way as in the Face Recognition test. The recognition score is ranged from -15 to 15. A higher score indicated a better visual, verbal long term memory.
Berg Balance Scale (BBS) | Baseline (0 week)
  The functional balance ability is measured by BBS. The BBS is an ordinal scale with 14 items, each item ranged from 0-4 with a total score ranged from 0-56. The higher score indicates a better balance function. Previous study has shown that BBS has good to excellent test-retest reliability (ICC=0.77-0.886) in older adults.
Berg Balance Scale (BBS) | Mid-intervention (5 week)
  The functional balance ability is measured by BBS. The BBS is an ordinal scale with 14 items, each item ranged from 0-4 with a total score ranged from 0-56. The higher score indicates a better balance function. Previous study has shown that BBS has good to excellent test-retest reliability (ICC=0.77-0.886) in older adults.
Berg Balance Scale (BBS) | Post-intervention (10 week)
  The functional balance ability is measured by BBS. The BBS is an ordinal scale with 14 items, each item ranged from 0-4 with a total score ranged from 0-56. The higher score indicates a better balance function. Previous study has shown that BBS has good to excellent test-retest reliability (ICC=0.77-0.886) in older adults.
Berg Balance Scale (BBS) | 1 month follow-up (14 week)
  The functional balance ability is measured by BBS. The BBS is an ordinal scale with 14 items, each item ranged from 0-4 with a total score ranged from 0-56. The higher score indicates a better balance function. Previous study has shown that BBS has good to excellent test-retest reliability (ICC=0.77-0.886) in older adults.
10 Meter Walking Test (10MWT) | Baseline (0 week)
  The walking speed over a short distance is measured by the 10MWT. The subject will be asked to walk 10 meter in a normal comfortable speed and maximum speed condition, respectively. The completion time will be records by stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged. The shorter the completion time, the better performance is. 10MWT has shown excellent test-retest reliability (ICC=0.98) in assessing healthy older adults.
10 Meter Walking Test (10MWT) | Mid-intervention (5 week)
  The walking speed over a short distance is measured by the 10MWT. The subject will be asked to walk 10 meter in a normal comfortable speed and maximum speed condition, respectively. The completion time will be records by stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged. The shorter the completion time, the better performance is. 10MWT has shown excellent test-retest reliability (ICC=0.98) in assessing healthy older adults.
10 Meter Walking Test (10MWT) | Post-intervention (10 week)
  The walking speed over a short distance is measured by the 10MWT. The subject will be asked to walk 10 meter in a normal comfortable speed and maximum speed condition, respectively. The completion time will be records by stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged. The shorter the completion time, the better performance is. 10MWT has shown excellent test-retest reliability (ICC=0.98) in assessing healthy older adults.
10 Meter Walking Test (10MWT) | 1 month follow-up (14 week)
  The walking speed over a short distance is measured by the 10MWT. The subject will be asked to walk 10 meter in a normal comfortable speed and maximum speed condition, respectively. The completion time will be records by stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged. The shorter the completion time, the better performance is. 10MWT has shown excellent test-retest reliability (ICC=0.98) in assessing healthy older adults.
6 Minutes Walking Test (6MWT) | Baseline (0 week)
  The aerobic capacity and walking endurance is measured by the 6MWT. The participants will be asked to walk as far as possible for 6 minutes in the 20 meters' corridor. The walking distance in 6 minutes will be records. The longer distance the subject walk, the better endurance is. The 6MWT has shown excellent test-retest reliability (ICC=0.95) in assessing healthy older adults.
6 Minutes Walking Test (6MWT) | Mid-intervention (5 week)
  The aerobic capacity and walking endurance is measured by the 6MWT. The participants will be asked to walk as far as possible for 6 minutes in the 20 meters' corridor. The walking distance in 6 minutes will be records. The longer distance the subject walk, the better endurance is. The 6MWT has shown excellent test-retest reliability (ICC=0.95) in assessing healthy older adults.
6 Minutes Walking Test (6MWT) | Post-intervention (10 week)
  The aerobic capacity and walking endurance is measured by the 6MWT. The participants will be asked to walk as far as possible for 6 minutes in the 20 meters' corridor. The walking distance in 6 minutes will be records. The longer distance the subject walk, the better endurance is. The 6MWT has shown excellent test-retest reliability (ICC=0.95) in assessing healthy older adults.
6 Minutes Walking Test (6MWT) | 1 month follow-up (14 week)
  The aerobic capacity and walking endurance is measured by the 6MWT. The participants will be asked to walk as far as possible for 6 minutes in the 20 meters' corridor. The walking distance in 6 minutes will be records. The longer distance the subject walk, the better endurance is. The 6MWT has shown excellent test-retest reliability (ICC=0.95) in assessing healthy older adults.
Time Up and Go Test (TUG) | Baseline (0 week)
  The functional ability is measured by TUG. The subject will be asked to stand up from the chair, walk 3 meters, turn 180°, go back to the chair and then sit down. The completion time will be recorded. The subjects need to repeat the test for 2 times. The completion time of the 2 trials will be averaged.
Time Up and Go Test (TUG) | Mid-intervention (5 week)
  The functional ability is measured by TUG. The subject will be asked to stand up from the chair, walk 3 meters, turn 180°, go back to the chair and then sit down. The completion time will be recorded. The subjects need to repeat the test for 2 times. The completion time of the 2 trials will be averaged.
Time Up and Go Test (TUG) | Post-intervention (10 week)
  The functional ability is measured by TUG. The subject will be asked to stand up from the chair, walk 3 meters, turn 180°, go back to the chair and then sit down. The completion time will be recorded. The subjects need to repeat the test for 2 times. The completion time of the 2 trials will be averaged.
Time Up and Go Test (TUG) | 1 month follow-up (14 week)
  The functional ability is measured by TUG. The subject will be asked to stand up from the chair, walk 3 meters, turn 180°, go back to the chair and then sit down. The completion time will be recorded. The subjects need to repeat the test for 2 times. The completion time of the 2 trials will be averaged.
Community Integration Measure | Baseline (0 week)
  The level of community integration is assessed by Chinese version of Community Integration Measure (CIM). It is a self-report questionnaire that is easily administrated to assess the community integration level. The instrument consists of 10 items, each rated from 1 to 5, giving a total score ranging from 10 to 50. A higher score indicates greater community integration. Liu et al. (Liu et al., 2014) reports that the Chinese version of the CIM showed good test-retest reliability (ICC=0.84) in people with stroke. A pilot study with 123 people with chronic stroke conducted as part of this research showed that CIM scores were significantly correlated with peak wrist flexion torque (r=0.203, p<0.05), Wolf Motoro Function Test (WMFT) scores (r=0.194, p<0.05) and Barthel Index scores (r=0.194, p<0.05).
Community Integration Measure | Mid-intervention (5 week)
  The level of community integration is assessed by Chinese version of Community Integration Measure (CIM). It is a self-report questionnaire that is easily administrated to assess the community integration level. The instrument consists of 10 items, each rated from 1 to 5, giving a total score ranging from 10 to 50. A higher score indicates greater community integration. Liu et al. reports that the Chinese version of the CIM showed good test-retest reliability (ICC=0.84) in people with stroke. A pilot study with 123 people with chronic stroke conducted as part of this research showed that CIM scores were significantly correlated with peak wrist flexion torque (r=0.203, p<0.05), WMFT scores (r=0.194, p<0.05) and Barthel Index scores (r=0.194, p<0.05).
Community Integration Measure | Post-intervention (10 week)
  The level of community integration is assessed by Chinese version of Community Integration Measure (CIM). It is a self-report questionnaire that is easily administrated to assess the community integration level. The instrument consists of 10 items, each rated from 1 to 5, giving a total score ranging from 10 to 50. A higher score indicates greater community integration. Liu et al. reports that the Chinese version of the CIM showed good test-retest reliability (ICC=0.84) in people with stroke. A pilot study with 123 people with chronic stroke conducted as part of this research showed that CIM scores were significantly correlated with peak wrist flexion torque (r=0.203, p<0.05), WMFT scores (r=0.194, p<0.05) and Barthel Index scores (r=0.194, p<0.05).
Community Integration Measure | 1 month follow-up (14 week)
  The level of community integration is assessed by Chinese version of Community Integration Measure (CIM). It is a self-report questionnaire that is easily administrated to assess the community integration level. The instrument consists of 10 items, each rated from 1 to 5, giving a total score ranging from 10 to 50. A higher score indicates greater community integration. Liu et al. reports that the Chinese version of the CIM showed good test-retest reliability (ICC=0.84) in people with stroke. A pilot study with 123 people with chronic stroke conducted as part of this research showed that CIM scores were significantly correlated with peak wrist flexion torque (r=0.203, p<0.05), WMFT scores (r=0.194, p<0.05) and Barthel Index scores (r=0.194, p<0.05).
Limit of Stability (LOS)-Reaction Time | Baseline (0 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Reaction time (RT) is used to assess the time participants take to give a movement response after cues are provided. The RT (second) in the 8 direction will be measured. The longer RT indicated poorer balance performance.
Limit of Stability (LOS)-Reaction Time | Mid-intervention (5 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Reaction time (RT) is used to assess the time participants take to give a movement response after cues are provided. The RT (second) in the 8 direction will be measured. The longer RT indicated poorer balance performance.
Limit of Stability (LOS)-Reaction Time | Post-intervention (10 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Reaction time (RT) is used to assess the time participants take to give a movement response after cues are provided. The RT (second) in the 8 direction will be measured. The longer RT indicated poorer balance performance.
Limit of Stability (LOS)-Reaction Time | 1 month follow-up (14 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Reaction time (RT) is used to assess the time participants take to give a movement response after cues are provided. The RT (second) in the 8 direction will be measured. The longer RT indicated poorer balance performance.
Limit of Stability (LOS)-Movement Velocity | Baseline (0 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Movement velocity (MV) is used to assess the average center of gravity (COG) displacement speed. The MV (degree/second) in the 8 direction will be measured. The smaller MV indicated poorer balance performance.
Limit of Stability (LOS)-Movement Velocity | Mid-intervention (5 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Movement velocity (MV) is used to assess the average center of gravity (COG) displacement speed. The MV (degree/second) in the 8 direction will be measured. The smaller MV indicated poorer balance performance.
Limit of Stability (LOS)-Movement Velocity | Post-intervention (10 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Movement velocity (MV) is used to assess the average center of gravity (COG) displacement speed. The MV (degree/second) in the 8 direction will be measured. The smaller MV indicated poorer balance performance.
Limit of Stability (LOS)-Movement Velocity | 1 month follow-up (14 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Movement velocity (MV) is used to assess the average center of gravity (COG) displacement speed. The MV (degree/second) in the 8 direction will be measured. The smaller MV indicated poorer balance performance.
Limit of Stability (LOS)-Endpoint Excursion | Baseline (0 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Endpoint excursion (EE) is used to assess how far the patient leans towards the target on his or her first attempt. The EE (%) in the 8 direction will be measured. The smaller EE indicated poorer balance performance.
Limit of Stability (LOS)-Endpoint Excursion | Mid-intervention (5 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Endpoint excursion (EE) is used to assess how far the patient leans towards the target on his or her first attempt. The EE (%) in the 8 direction will be measured. The smaller EE indicated poorer balance performance.
Limit of Stability (LOS)-Endpoint Excursion | Post-intervention (10 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Endpoint excursion (EE) is used to assess how far the patient leans towards the target on his or her first attempt. The EE (%) in the 8 direction will be measured. The smaller EE indicated poorer balance performance.
Limit of Stability (LOS)-Endpoint Excursion | 1 month follow-up (14 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Endpoint excursion (EE) is used to assess how far the patient leans towards the target on his or her first attempt. The EE (%) in the 8 direction will be measured. The smaller EE indicated poorer balance performance.
Limit of Stability (LOS)-Maximum Excursion | Baseline (0 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Maximum excursion (ME) is used to assess the maximum amount the patient leaned during the trial. The ME (%) in the 8 direction will be measured. The smaller ME indicated poorer balance performance.
Limit of Stability (LOS)-Maximum Excursion | Mid-intervention (5 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Maximum excursion (ME) is used to assess the maximum amount the patient leaned during the trial. The ME (%) in the 8 direction will be measured. The smaller ME indicated poorer balance performance.
Limit of Stability (LOS)-Maximum Excursion | Post-intervention (10 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Maximum excursion (ME) is used to assess the maximum amount the patient leaned during the trial. The ME (%) in the 8 direction will be measured. The smaller ME indicated poorer balance performance.
Limit of Stability (LOS)-Maximum Excursion | 1 month follow-up (14 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Maximum excursion (ME) is used to assess the maximum amount the patient leaned during the trial. The ME (%) in the 8 direction will be measured. The smaller ME indicated poorer balance performance.
Limit of Stability (LOS)-Directional Control | Baseline (0 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Directional control (DC) is used to assess how much of the patient's movement was in the target direction. The DC (%) in the 8 direction will be measured. The smaller DC indicated poorer balance performance.
Limit of Stability (LOS)-Directional Control | Mid-intervention (5 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Directional control (DC) is used to assess how much of the patient's movement was in the target direction. The DC (%) in the 8 direction will be measured. The smaller DC indicated poorer balance performance.
Limit of Stability (LOS)-Directional Control | Post-intervention (10 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Directional control (DC) is used to assess how much of the patient's movement was in the target direction. The DC (%) in the 8 direction will be measured. The smaller DC indicated poorer balance performance.
Limit of Stability (LOS)-Directional Control | 1 month follow-up (14 week)
  The LOS is measured by the balance plate system (Bertec, Columbus, OH). During the limits of stability task, subjects were instructed to shift their weight by moving their pelvis and torso without flexing their hips or knees, keeping their heels in contact with the force plates and their arms/hands at their sides. The subjects will be instructed to shifted his or her center of mass to forward (0°), right-forward (45°), right (90°), right-backward (135°), backward (180°), left backward (225°), left (270°) and left-forward (315°), based on a visual projection of the center of mass in the current and target locations. The duration of each weight shifting trial was 10 seconds. Directional control (DC) is used to assess how much of the patient's movement was in the target direction. The DC (%) in the 8 direction will be measured. The smaller DC indicated poorer balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Shamay Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Alzheimer's Association. 2015 Alzheimer's disease facts and figures. Alzheimers Dement. 2015 Mar;11(3):332-84. doi: 10.1016/j.jalz.2015.02.003. PMID 25984581
- [Background] Beste C, Steenbergen L, Sellaro R, Grigoriadou S, Zhang R, Chmielewski W, Stock AK, Colzato L. Effects of Concomitant Stimulation of the GABAergic and Norepinephrine System on Inhibitory Control - A Study Using Transcutaneous Vagus Nerve Stimulation. Brain Stimul. 2016 Nov-Dec;9(6):811-818. doi: 10.1016/j.brs.2016.07.004. Epub 2016 Jul 19. PMID 27522167
- [Background] Burger AM, Verkuil B, Van Diest I, Van der Does W, Thayer JF, Brosschot JF. The effects of transcutaneous vagus nerve stimulation on conditioned fear extinction in humans. Neurobiol Learn Mem. 2016 Jul;132:49-56. doi: 10.1016/j.nlm.2016.05.007. Epub 2016 May 21. PMID 27222436
- [Background] Elwood RW. The Wechsler Memory Scale-Revised: psychometric characteristics and clinical application. Neuropsychol Rev. 1991 Jun;2(2):179-201. doi: 10.1007/BF01109053. PMID 1844708
- [Background] Gates NJ, Rutjes AW, Di Nisio M, Karim S, Chong LY, March E, Martinez G, Vernooij RW. Computerised cognitive training for 12 or more weeks for maintaining cognitive function in cognitively healthy people in late life. Cochrane Database Syst Rev. 2020 Feb 27;2(2):CD012277. doi: 10.1002/14651858.CD012277.pub3. PMID 32104914
- [Background] Hein E, Nowak M, Kiess O, Biermann T, Bayerlein K, Kornhuber J, Kraus T. Auricular transcutaneous electrical nerve stimulation in depressed patients: a randomized controlled pilot study. J Neural Transm (Vienna). 2013 May;120(5):821-7. doi: 10.1007/s00702-012-0908-6. Epub 2012 Nov 2. PMID 23117749
- [Background] Hiengkaew V, Jitaree K, Chaiyawat P. Minimal detectable changes of the Berg Balance Scale, Fugl-Meyer Assessment Scale, Timed "Up & Go" Test, gait speeds, and 2-minute walk test in individuals with chronic stroke with different degrees of ankle plantarflexor tone. Arch Phys Med Rehabil. 2012 Jul;93(7):1201-8. doi: 10.1016/j.apmr.2012.01.014. Epub 2012 Apr 12. PMID 22502805
- [Background] Holbein-Jenny MA, Billek-Sawhney B, Beckman E, Smith T. Balance in personal care home residents: a comparison of the Berg Balance Scale, the Multi-Directional Reach Test, and the Activities-Specific Balance Confidence Scale. J Geriatr Phys Ther. 2005;28(2):48-53. PMID 16236228
- [Background] Jansen WJ, Ossenkoppele R, Knol DL, Tijms BM, Scheltens P, Verhey FR, Visser PJ; Amyloid Biomarker Study Group; Aalten P, Aarsland D, Alcolea D, Alexander M, Almdahl IS, Arnold SE, Baldeiras I, Barthel H, van Berckel BN, Bibeau K, Blennow K, Brooks DJ, van Buchem MA, Camus V, Cavedo E, Chen K, Chetelat G, Cohen AD, Drzezga A, Engelborghs S, Fagan AM, Fladby T, Fleisher AS, van der Flier WM, Ford L, Forster S, Fortea J, Foskett N, Frederiksen KS, Freund-Levi Y, Frisoni GB, Froelich L, Gabryelewicz T, Gill KD, Gkatzima O, Gomez-Tortosa E, Gordon MF, Grimmer T, Hampel H, Hausner L, Hellwig S, Herukka SK, Hildebrandt H, Ishihara L, Ivanoiu A, Jagust WJ, Johannsen P, Kandimalla R, Kapaki E, Klimkowicz-Mrowiec A, Klunk WE, Kohler S, Koglin N, Kornhuber J, Kramberger MG, Van Laere K, Landau SM, Lee DY, de Leon M, Lisetti V, Lleo A, Madsen K, Maier W, Marcusson J, Mattsson N, de Mendonca A, Meulenbroek O, Meyer PT, Mintun MA, Mok V, Molinuevo JL, Mollergard HM, Morris JC, Mroczko B, Van der Mussele S, Na DL, Newberg A, Nordberg A, Nordlund A, Novak GP, Paraskevas GP, Parnetti L, Perera G, Peters O, Popp J, Prabhakar S, Rabinovici GD, Ramakers IH, Rami L, Resende de Oliveira C, Rinne JO, Rodrigue KM, Rodriguez-Rodriguez E, Roe CM, Rot U, Rowe CC, Ruther E, Sabri O, Sanchez-Juan P, Santana I, Sarazin M, Schroder J, Schutte C, Seo SW, Soetewey F, Soininen H, Spiru L, Struyfs H, Teunissen CE, Tsolaki M, Vandenberghe R, Verbeek MM, Villemagne VL, Vos SJ, van Waalwijk van Doorn LJ, Waldemar G, Wallin A, Wallin AK, Wiltfang J, Wolk DA, Zboch M, Zetterberg H. Prevalence of cerebral amyloid pathology in persons without dementia: a meta-analysis. JAMA. 2015 May 19;313(19):1924-38. doi: 10.1001/jama.2015.4668. PMID 25988462
- [Background] Jonsdottir S, Bouma A, Sergeant JA, Scherder EJ. Effects of transcutaneous electrical nerve stimulation (TENS) on cognition, behavior, and the rest-activity rhythm in children with attention deficit hyperactivity disorder, combined type. Neurorehabil Neural Repair. 2004 Dec;18(4):212-21. doi: 10.1177/1545968304270759. PMID 15537992
- [Background] Langa KM, Levine DA. The diagnosis and management of mild cognitive impairment: a clinical review. JAMA. 2014 Dec 17;312(23):2551-61. doi: 10.1001/jama.2014.13806. PMID 25514304
- [Background] Liu TW, Ng SS, Ng GY. Translation and initial validation of the Chinese (Cantonese) version of community integration measure for use in patients with chronic stroke. Biomed Res Int. 2014;2014:623836. doi: 10.1155/2014/623836. Epub 2014 Jun 4. PMID 24995317
- [Background] Luijpen MW, Swaab DF, Sergeant JA, van Dijk KR, Scherder EJ. Effects of transcutaneous electrical nerve stimulation (TENS) on memory in elderly with mild cognitive impairment. Behav Brain Res. 2005 Mar 30;158(2):349-57. doi: 10.1016/j.bbr.2004.09.017. PMID 15698902
- [Background] Prince, M. J., Wimo, A., Guerchet, M. M., Ali, G. C., Wu, Y. T., & Prina, M. (2015). World Alzheimer Report 2015-The Global Impact of Dementia: An analysis of prevalence, incidence, cost and trends.
- [Background] Scherder EJ, Bouma A. Effects of transcutaneous electrical nerve stimulation on memory and behavior in Alzheimer's disease may be stage-dependent. Biol Psychiatry. 1999 Mar 15;45(6):743-9. doi: 10.1016/s0006-3223(98)00072-9. PMID 10188004
- [Background] Scherder EJ, Bouma A, Steen L. Influence of transcutaneous electrical nerve stimulation on memory in patients with dementia of the Alzheimer type. J Clin Exp Neuropsychol. 1992 Nov;14(6):951-60. doi: 10.1080/01688639208402546. PMID 1360474
- [Background] Scherder EJ, Bouma A, Steen LM. Effects of "isolated" transcutaneous electrical nerve stimulation on memory and affective behavior in patients with probable Alzheimer's disease. Biol Psychiatry. 1998 Mar 15;43(6):417-24. doi: 10.1016/s0006-3223(97)00208-4. PMID 9532346
- [Background] Sellaro R, de Gelder B, Finisguerra A, Colzato LS. Transcutaneous vagus nerve stimulation (tVNS) enhances recognition of emotions in faces but not bodies. Cortex. 2018 Feb;99:213-223. doi: 10.1016/j.cortex.2017.11.007. Epub 2017 Nov 23. PMID 29275193
- [Background] Sellaro R, van Leusden JW, Tona KD, Verkuil B, Nieuwenhuis S, Colzato LS. Transcutaneous Vagus Nerve Stimulation Enhances Post-error Slowing. J Cogn Neurosci. 2015 Nov;27(11):2126-32. doi: 10.1162/jocn_a_00851. Epub 2015 Jul 30. PMID 26226074
- [Background] Shimada, Hiroyuki, Sangyoon Lee, and Hyuma Makizako.
- [Background] Shimada H, Makizako H, Doi T, Lee S, Lee S. Conversion and Reversion Rates in Japanese Older People With Mild Cognitive Impairment. J Am Med Dir Assoc. 2017 Sep 1;18(9):808.e1-808.e6. doi: 10.1016/j.jamda.2017.05.017. Epub 2017 Jul 12. PMID 28711424
- [Background] Steenbergen L, Sellaro R, Stock AK, Verkuil B, Beste C, Colzato LS. RETRACTED: Transcutaneous vagus nerve stimulation (tVNS) enhances response selection during action cascading processes. Eur Neuropsychopharmacol. 2015 Jun;25(6):773-8. doi: 10.1016/j.euroneuro.2015.03.015. Epub 2015 Mar 30. PMID 25869158
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Stroop, J. R. (1935). Studies of interference in serial verbal reactions. Journal of experimental psychology, 18(6), 643.
- [Background] Thomas KR, Edmonds EC, Eppig JS, Wong CG, Weigand AJ, Bangen KJ, Jak AJ, Delano-Wood L, Galasko DR, Salmon DP, Edland SD, Bondi MW; Alzheimer's Disease Neuroimaging Initiative. MCI-to-normal reversion using neuropsychological criteria in the Alzheimer's Disease Neuroimaging Initiative. Alzheimers Dement. 2019 Oct;15(10):1322-1332. doi: 10.1016/j.jalz.2019.06.4948. Epub 2019 Sep 5. PMID 31495605
- [Background] Viveiro LAP, Gomes GCV, Bacha JMR, Carvas Junior N, Kallas ME, Reis M, Jacob Filho W, Pompeu JE. Reliability, Validity, and Ability to Identity Fall Status of the Berg Balance Scale, Balance Evaluation Systems Test (BESTest), Mini-BESTest, and Brief-BESTest in Older Adults Who Live in Nursing Homes. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):E45-E54. doi: 10.1519/JPT.0000000000000215. PMID 30407272
- [Background] de Wall C, Wilson BA, Baddeley AD. The Extended Rivermead Behavioural Memory Test: a measure of everyday memory performance in normal adults. Memory. 1994 Jun;2(2):149-66. doi: 10.1080/09658219408258942. PMID 7584289
- [Background] Wang, R.-Y., Zhou, J.-H., Huang, Y.-C., & Yang, Y.-R. (2018). Reliability of the Chinese version of the Trail Making Test and Stroop Color and Word Test among older adults. International Journal of Gerontology, 12(4), 336-339.
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421